CLINICAL TRIAL: NCT04532645
Title: A Pan-European Non-interventional, Retrospective Observational Cohort Study of Patients With BRCA Mutated Advanced (FIGO Stage III-IV) Ovarian Cancer Treated With Olaparib Tablets in the First-line Maintenance Setting
Brief Title: Olaparib Real-world Utilization and Clinical Outcomes in France, Italy, and the UK
Acronym: OVAL-1
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00019
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Ovary Cancer
Keywords: Ovary cancer; Ovarian neoplasm; BRCA mutated advanced (FIGO stage III-IV) ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with BRCA mutated ovarian cancer: BRCA mutated advanced (FIGO stage III-IV) ovarian cancer patients who received first dose maintenance olaparib in 1L setting
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib
  Other Names: Lynparza

SUMMARY:
This is a retrospective observational medical records review study of BRCA mutated advanced (FIGO stage III-IV) ovarian cancer patients who received first dose maintenance olaparib in 1L setting in France, Italy and the UK. Physicians who treated ovarian cancer patients with olaparib in 1L setting will be requested to recruit patients to have their clinical data abstracted from their clinical records in line with local laws

DETAILED DESCRIPTION:
Primary Objective(s)

1. To estimate progression-free survival (PFS) in patients with BRCA-mutated advanced ovarian cancer treated with olaparib tablets in real-world first line maintenance setting.
2. To describe olaparib treatment patterns (dosage; frequency of: dosage changes, dose interruptions, treatment cessation) in patients with BRCA-mutated advanced ovarian cancer treated in real-world first line maintenance setting.

Secondary Objective(s)

1. To estimate overall survival (OS) in patients with BRCA-mutated advanced ovarian cancer treated with olaparib tablets in real-world first line maintenance setting.
2. To describe reasons for olaparib dosage changes, dose interruptions and treatment cessation in patients with BRCA-mutated advanced ovarian cancer treated in real-world first line maintenance setting
3. To describe surgical and chemotherapy outcomes (PR/CR) in patients with BRCA-mutated advanced ovarian cancer before initiation of real-world first line maintenance olaparib tablets
4. To describe response rate (RR) to olaparib tablets in patients with BRCA-mutated ovarian cancer with partial response to real-world first line chemotherapy.
5. To describe treatment patterns and clinical outcomes in patients with BRCA-mutated advanced ovarian cancer who progressed during olaparib real-world first line maintenance therapy (including frequency of treatment interruptions, dosage reductions and treatment discontinuations and reasons associated with patterns)
6. To estimate second progression-free survival (PFS2) in patients with BRCA-mutated ovarian cancer who progress while on olaparib real-world first line maintenance therapy.
7. To describe healthcare resource utilisation in patients with BRCA-mutated advanced ovarian cancer treated with olaparib in real-world first line setting

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, histologically confirmed, advanced (FIGO stage III - IV) epithelial ovarian cancer, primary peritoneal cancer and / or fallopian-tube cancer who have completed first line platinum-based chemotherapy, in PR/CR and treated with at least one dose of olaparib in first line maintenance setting
* Patients aged ≥18 years old
* Ability and/or willingness to provide a signed informed consent form (where required)

Exclusion Criteria:

* Withdrawal of informed consent (where consent required)
* Concurrent participation in any clinical study with an investigational product at the time of olaparib initiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Patients with BRCA mutated advanced (FIGO stage III-IV) ovarian cancer treated with olaparib in first-line maintenance setting
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Progression | 36 months
  Progression-free survival (PFS)

SECONDARY OUTCOMES:
Overall Survival | 36 months
  Overall survival over 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Gourley, MD, PhD, Principal Investigator — University of Edinburgh; Domenica Lorusso, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS; Delphine Garbay, MD, Principal Investigator — Institut Bergonie, France
Locations (49):
- France (19):
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Calais
  - Research Site, Chambray-lès-Tours
  - Research Site, Epagny Metz-Tessy
  - Research Site, Grenoble
  - Research Site, Langon
  - Research Site, Lyon
  - Research Site, Nancy
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Roubaix
  - Research Site, Saint-Cloud
  - Research Site, Saint-Grégoire
  - Research Site, Suresnes
  - Research Site, Tours
  - Research Site, Villejuif
- Italy (15):
  - Research Site, Acquaviva delle Fonti
  - Research Site, Aviano
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Cagliari
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Negrar
  - Research Site, Parma
  - Research Site, Roma
  - Research Site, Torino
- United Kingdom (15):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Ediburgh
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Manchester
  - Research Site, Newcastle
  - Research Site, Northampton
  - Research Site, Nottingham
  - Research Site, Portsmouth
  - Research Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: ICF, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0817R00019&attachmentIdentifier=340e7003-5eea-4823-ad07-0a1b9c2731ee&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=